CLINICAL TRIAL: NCT03242109
Title: An Epidemiological Study of Risk Factors for Cardiovascular Disease and Tumors in an Adult Population of the Molise Region
Brief Title: The Moli-sani Study
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, MD, PhD, Neuromed IRCCS
Other Study IDs: 50/17
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Cancer; Neurodegenerative Diseases; Diabetes; Pulmonary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Neurodegenerative Diseases; Diabetes Mellitus; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples obtained from participants who had fasted overnight and had refrained from smoking for at least 6 h and stored in liquid nitrogen in the Biological bank of the Moli-sani study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease and malignancies account for more than 70% of all causes of mortality and morbidity in Italy. There is a subtle balance between genetic determinants and lifestyle, that often defines the line between health and sickness. So far studies aiming at identifying risk factors have mainly come from Northern Europe and the USA. It was to understand this balance between genetics and environmental determinants better, and to tailor appropriate preventive strategies for Italian and other Southern European populations, that the Moli-sani study was launched, transforming a small Italian region into a large scientific laboratory: the "Molise lab".

Each participant received a thorough medical check-up at no cost to either him/her or the national health service, resulting in thousands of hours of free public health care. With a completely computerized system, Moli-sani is a "paperless" study, in which researchers and participants communicate using recently developed technologies such as mobile phone text messages (SMS). The biological data bank (the "MoliBank") is one of the largest in Europe. Paying particular attention towards innovation and new technologies, the Moli-sani study has placed itself at the cutting edge of a new paradigm crossing research and prevention

DETAILED DESCRIPTION:
The cohort of the Moli-sani study has recruited 24,325 persons, aged >35 years, resident in the Molise region.The latter covers an area of 4,438 Km2, including 136 towns. Participants are recruited from city-hall registries by a multistage sampling. Firstly townships were sampled in three major areas of Molise region, starting from the main cities (Campobasso, Termoli, Isernia) by cluster sampling, then, within each township, participants are selected by simple random sampling, using electronically generated numbers.Exclusion criteria are pregnancy at the time of recruitment, disturbances in understanding or willingness, current poly-traumas or coma, refusal to sign the Informed Consent form. All subjects identified are sent a letter inviting them to participate in the project, followed a few days later by a phone call. The recruitment started in the area of Campobasso, then it moved to the areas of Termoli.

ELIGIBILITY:
Inclusion Criteria:

* Resident in the Molise region (Italy), aged >35.

Exclusion Criteria:

* pregnancy at the time of recruitment, disturbances in understanding or willingness, current poly-traumas or coma, refusal to sign the Informed Consent form.

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Moli-sani is a population-based cohort study that recruited, between March 2005 and April 2010, 24,325 men and women at random from individuals aged 35 years or older resident in the Molise region, to investigate genetic and environmental risk factors for cardiovascular, cerebrovascular and tumour diseases.
Sampling Method: Probability Sample
Enrollment: 24325 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2010-04-30 (Actual); Study Completion 2010-04-30 (Actual)

PRIMARY OUTCOMES:
Primary cardiovascular diseases | 10 years
  Primary fatal and nonfatal incident cases of CHD (unstable angina, myocardial infarction, coronary revascularization and sudden death for unspecified cardiac event) and cerebrovascular disease that occurred in the cohort during follow-up
Cancer | 10 years
  Primary fatal and nonfatal incident cases of cancer that occurred in the cohort during follow-up, assessed by cross-linkage with hospital discharge record and regional death registry
Heart failure | 10 years
  Primary fatal and nonfatal incident cases of heart failure that occurred in the cohort during follow-up, assessed by cross-linkage with hospital discharge record and regional death registry
Atrial fibrillation | 10 years
  Primary fatal and nonfatal incident cases of atrial fibrillation that occurred in the cohort during follow-up, assessed by cross-linkage with hospital discharge record and regional death registry
Diabetes | 10 years
  Primary incident cases of diabetes that occurred in the cohort during follow-up, assessed by cross-linkage with hospital discharge record and regional death registry or pharmacological prescription registry. Diabetes onset is defined as blood glucose ≥126 mg/dl or by use of specific pharmacological treatment

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, MD, PhD, Principal Investigator — Department of Epidemiology and Prevention, IRCCS Neuromed
Locations (1):
- Irccs Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: Yes
sumbmission of a research proposal form to be approved by the Moli-sani scientific committee and signature of a research agreement.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Upon request
Access Criteria: Approval by the Moli-sani study Scientific committee

REFERENCES:
- [Result] Pounis G, Tabolacci C, Costanzo S, Cordella M, Bonaccio M, Rago L, D'Arcangelo D, Filippo Di Castelnuovo A, de Gaetano G, Donati MB, Iacoviello L, Facchiano F; Moli-sani study investigators. Reduction by coffee consumption of prostate cancer risk: Evidence from the Moli-sani cohort and cellular models. Int J Cancer. 2017 Jul 1;141(1):72-82. doi: 10.1002/ijc.30720. Epub 2017 Apr 24. PMID 28436066
- [Result] Bonaccio M, Di Castelnuovo A, Costanzo S, de Curtis A, Persichillo M, Cerletti C, Donati MB, de Gaetano G, Iacoviello L; MOLI-SANI study Investigators. Mean platelet volume is associated with lower risk of overall and non-vascular mortality in a general population. Results from the Moli-sani study. Thromb Haemost. 2017 Jun 2;117(6):1129-1140. doi: 10.1160/TH16-12-0974. Epub 2017 Mar 30. PMID 28357442